CLINICAL TRIAL: NCT06178835
Title: Erythropoietin for the Prevention of Postoperative Delirium in Elderly Patients Undergoing Total Joint Arthroplasty: Randomized Controlled Study
Brief Title: EPO for Postop Delirium in Elderly Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 4-2017-0694
Record Dates: First submitted 2023-12-12; First posted 2023-12-21 (Actual); Last update posted 2023-12-21 (Actual); Status verified 2023-12

CONDITIONS: Postoperative Delirium
MeSH Terms: conditions — Emergence Delirium | interventions — Erythropoietin; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Erythropoietin (Experimental): 500 IU/kg of EPO given intramuscularly 3 times for each patient
  Interventions: Drug: Erythropoietin
- Control (Placebo Comparator): Same amount of normal saline given intramuscularly 3 times for each patient
  Interventions: Drug: normal saline

INTERVENTIONS:
Drug: Erythropoietin — 500 IU/kg of erythropoietin is given 3 times for each patient: the day before surgery, start of surgery and on postoperative day 1.
  Arms: Erythropoietin
Drug: normal saline — The same amount of normal saline is given 3 times for each patient: the day before surgery, start of surgery and on postoperative day 1.
  Arms: Control

SUMMARY:
Postoperative delirium is a common complication after surgery. The underlying pathophysiology of this complication is unclear, however neuroinflammation and oxidative stress secondary to surgery had shown to be the cause of postoperative cognitive dysfunction and delirium. Erythropoietin represents non-erythropoietic effects of anti-inflammatory properties. The aims of this study were to determine the role of erythropoietin toward the development of postoperative delirium, in terms of changes in inflammatory reaction by affecting the innate immunity in elderly patients undergoing total joint arthroplasty surgery.

ELIGIBILITY:
Inclusion Criteria:

* Age 65 years and older
* Patients scheduled for elective total knee arthroplasty, total hip arthroplasty

Exclusion Criteria:

* Unable to communicate
* Cognitive impairment
* Unable to pre-screen delirium due to underlying central nervous system disease
* History of hypersensitivity related to erythropoietin and other anesthesia-related drugs
* History of myocardial infarction, pulmonary infarction, cerebral infarction, ischemic vascular disease, epilpesy, chronic liver disease, chronic kidney disease
* Uncontrolled high blood pressure
* Within one month of starting anti-hypertensive medication

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 76 (Actual)
Dates: Start 2017-09-12 (Actual); Primary Completion 2019-07-28 (Actual); Study Completion 2019-08-28 (Actual)

PRIMARY OUTCOMES:
Incidence of delirium | 2 days post surgery, 5 days post surgery
  Development of postoperative delirium determined by validated evaluation tests.

SECONDARY OUTCOMES:
Inflammatory biomarker | before surgery, after surgery, 3 days post surgery day 3
  Preoperative and postoperative comparison of inflammatory biomarkers (IL-1, IL-6, TNF-a)

CONTACTS AND LOCATIONS:
Overall Officials: Bon-Nyeo Koo, Principal Investigator — Department of Anesthesiology and Pain medicine, Severance Hospital, Seoul, South Korea
Locations (1):
- Department of Anesthesiology and Pain medicine, Severance Hospital, Seoul, South Korea, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kim EJ, Park KK, Choi SY, Ju HM, Kim TL, Kim J, Kim SY, Koo BN. Erythropoietin for the prevention of postoperative neurocognitive disorder in older adult patients undergoing total joint arthroplasty: a randomized controlled study. BMC Anesthesiol. 2024 Nov 15;24(1):418. doi: 10.1186/s12871-024-02770-9. PMID 39548414